CLINICAL TRIAL: NCT04233073
Title: Prospective, Open-Label Clinical Study of Andexanet Alfa in Patients Receiving FXa (Activated Factor X) Inhibitor Who Require Urgent Surgery
Brief Title: Trial of Andexanet in Patients Receiving an Oral FXa Inhibitor Who Require Urgent Surgery
Acronym: Annexa-S
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Limited value as a single-arm study
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALXN2070-19-515
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-02

CONDITIONS: Surgery
Keywords: Urgent Surgery; Thrombosis; Anticoagulant; Surgery; Surgical; Abdominal; Thoracic; Orthopedic; Gynecological; Laparoscopic; Neurosurgery; Gastrointestinal
MeSH Terms: conditions — Thrombosis | interventions — PRT064445

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: andexanet alfa — Andexanet is a recombinant version of human FXa
  Other Names: Andexxa®; Ondexxya®

SUMMARY:
Prospective, open-label clinical trial to evaluate the efficacy and safety of andexanet alfa patients who require urgent surgery that have been anticoagulated with the FXa (activated factor X) inhibitors.

DETAILED DESCRIPTION:
This is a multicenter, prospective, open-label study to determine the efficacy and safety of andexanet in patients who require urgent surgery who have received 1 of the following FXa inhibitors: apixaban, rivaroxaban, edoxaban, or enoxaparin. The start of surgery must be within 15 hours following the last dose of FXa inhibitor. The primary efficacy outcome will be adjudicated by an independent Endpoint Adjudication Committee.

ELIGIBILITY:
Inclusion Criteria:

All of the following criteria must be met for the patient to be eligible:

* Either the patient or their medical proxy (or legal designee) has given written informed consent.
* Age ≥ 18 and < 85 years old.
* Requires urgent surgical intervention that must occur within 12 hours of consent, for which reversal of anti-fXa activity is judged necessary.
* Treatment with an oral FXa inhibitor (apixaban [last dose 2.5 mg or greater], rivaroxaban [last dose 10 mg or greater], edoxaban [last dose 30 mg or greater] or enoxaparin [≥ 1 mg/kg/d]):
* ≤ 15 hours prior to start of surgery.
* > 15 hours prior to start of surgery or unknown time from the last dose, if documented anti fXa activity is > 100 ng/mL (> 0.5 IU/mL for enoxaparin, or over the equivalent IU/mL threshold on a low molecular weight heparin assay; see Laboratory Manual) within 2 hours prior to consent. Note: Patients enrolled in this manner should receive a high-andexanet dosing regimen.
* Have a negative pregnancy test documented prior to enrollment (for women of childbearing potential).
* Willingness to use highly effective methods of contraception through 30 days following study drug dose (for female and male patients who are fertile).

Exclusion Criteria:

If a patient meets any of the following criteria, he or she is not eligible:

* Surgery for which the risk of clinically meaningful uncontrolled or unmanageable bleeding is low.
* Acute life-threatening bleeding (ISTH criteria) at the time of Screening:

  1. The patient has acute-overt bleeding that is potentially life-threatening, e.g., with signs or symptoms of hemodynamic compromise, such as severe hypotension, poor skin perfusion, mental confusion, low urine output that cannot be otherwise explained.
  2. The patient has overt bleeding associated with a fall in hemoglobin level by ≥2g/dL, OR, a hemoglobin ≤8 g/dL if no baseline hemoglobin is available.
  3. The patient has acute bleeding in a critical area or organ, such as pericardial, intracranial, or intraspinal.
* Any surgical procedure that involves the intraoperative use of systemic, intravascular, unfractionated heparin.
* Primary procedure for efficacy assessment is a non-surgical interventional procedure (e.g, lumbar puncture, skin biopsy, cardiac catheterization, endoscopic retrograde cholangio-pancreatography).
* Expected survival of < 1 month due to comorbidity.
* Known "Do Not Resuscitate" order or similar advanced directive.
* The patient has a recent history (within 30 days prior to screening) of a diagnosed TE as follows: venous thromboembolism (including deep vein thrombosis, pulmonary embolism, intracardiac thrombus), myocardial infarction (including asymptomatic troponin elevations), disseminated intravascular coagulation, acute traumatic coagulopathy, cerebrovascular accident, transient ischemic attack, unstable angina pectoris hospitalization, or severe peripheral vascular disease.
* Acute decompensated heart failure or cardiogenic shock at the time of screening.
* The patient has sepsis or septic or severe hemorrhagic shock at the time of Screening.
* The patient has heparin-induced thrombocytopenia (with or without thrombosis).
* Inherited coagulopathy (e.g., anti-phospholipid antibody syndrome, protein C/S deficiency, Factor V Leiden) at time of Screening.
* Platelet count < 80,000/µL at the time of Screening.
* Last dose of apixaban < 2.5 mg, rivaroxaban < 10 mg, edoxaban < 30 mg, or enoxaparin 40 mg.
* The patient is pregnant or a lactating female.
* The patient has received any of the following drugs or blood products within 7 days of enrollment:

  * Vitamin K antagonists (e.g., warfarin).
  * Dabigatran.
  * Prothrombin complex concentrate products (e.g., Kcentra®) or recombinant factor VIIa (e.g., NovoSeven®).
  * Whole blood, plasma fractions. Note: Administration of tranexamic acid, platelets or packed red blood cells is not an exclusion criterion.
* The patient was treated with an investigational drug < 30 days prior to Screening.
* Prior treatment with andexanet.
* Known hypersensitivity to any component of andexanet.
* Known allergic reaction to hamster proteins.
* Known or suspected (i.e., presumed positive) COVID-19-related illness at the time of Screening.

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-27 (Actual); Primary Completion 2021-11-23 (Actual); Study Completion 2022-01-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (51):
- United States (18):
  - Clinical Trial Site, Phoenix, Arizona
  - Clinical Trial Site, Tucson, Arizona
  - Clinical Trial Site, Long Beach, California
  - Clinical Trial Site, Moreno Valley, California
  - Clinical Trial Site, Washington D.C., District of Columbia
  - Clinical Trial Site, Sarasota, Florida
  - Clinical Trial Site, Tampa, Florida
  - Clinical Trial Site, Iowa City, Iowa
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, Camden, New Jersey
  - Clinical Trial Site, Staten Island, New York
  - Clinical Trial Site, Charlotte, North Carolina
  - Clinical Trial Site, Durham, North Carolina
  - Clinical Trial Site, Columbus, Ohio
  - Clinical Trial Site, Tulsa, Oklahoma
  - Clinical Trial Site, Portland, Oregon
  - Clinical Trial Site, Philadelphia, Pennsylvania
  - Clinical Trial Site, Pittsburgh, Pennsylvania
- Austria (4):
  - Clinical Trial Site, Graz
  - Clinical Trial Site, Innsbruck
  - Clinical Trial Site, Klagenfurt
  - Clinical Trial Site, Vienna
- France (5):
  - Clinical Trial Site, Clermont-Ferrand
  - Clinical Trial Site, Dijon
  - Clinical Trial Site, Lille
  - Clinical Trial Site, Nantes
  - Clinical Trial Site, Paris
- Germany (11):
  - Clinical Trial Site, Aachen
  - Clinical Trial Site, Bonn
  - Clinical Trial Site, Cologne
  - Clinical Trial Site, Dortmund
  - Clinical Trial Site, Freiburg im Breisgau
  - Clinical Trial Site, Giessen
  - Clinical Trial Site, Heidelberg
  - Clinical Trial Site, Konstanz
  - Clinical Trial Site, Mainz
  - Clinical Trial Site, Murnau am Staffelsee
  - Clinical Trial Site, Würzburg
- Israel (4):
  - Clinical Trial Site, Ashkelon
  - Clinical Trial Site, Haifa
  - Clinical Trial Site, Jerusalem
  - Clinical Trial Site, Petah Tikva
- Japan (9):
  - Clinical Trial Site, Kamakura
  - Clinical Trial Site, Kasuga
  - Clinical Trial Site, Kawasaki
  - Clinical Trial Site, Kumamoto
  - Clinical Trial Site, Kurume
  - Clinical Trial Site, Nagoya
  - Clinical Trial Site, Sakai
  - Clinical Trial Site, Sendai
  - Clinical Trial Site, Tokyo

IPD SHARING:
Plan to Share IPD: Yes
Alexion has a public commitment to allow requests for access to study data and will be supplying a protocol, CSR, and plain language summaries.
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- [Derived] Levy JH, Mamoun N. Direct oral anticoagulants and their antagonists in perioperative practice. Curr Opin Anaesthesiol. 2023 Aug 1;36(4):394-398. doi: 10.1097/ACO.0000000000001275. Epub 2023 Jun 6. PMID 37314165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who required urgent surgery and received factor Xa (fXa) inhibitors (apixaban, rivaroxaban, edoxaban, or enoxaparin) before surgery were enrolled in the study.
Pre-assignment Details: This study is a single-arm study and all participants received 1 of 2 doses of andexanet based on the specific anticoagulant taken. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Groups:
- Andexanet Alfa: Participants received a dose of andexanet alfa based on the specific FXa inhibitor, dose, and time since the last dose (<8 hours, ≥8 hours, or unknown).
Period: Overall Study
Arm/Group | Andexanet Alfa
Started | 10
Treated With Any Amount of Andexanet | 10
Efficacy Set | 6
Completed | 5
Not Completed | 5
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Population: Safety Set: Participants who were enrolled into the study and treated with any amount of andexanet alfa. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Arm/Group | Andexanet Alfa
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: Years] | 79.8 [68 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per local law, ethnicity data not collected for participants located in France.
  Participants
    number analyzed (Participants) | 6
    Hispanic or Latino | 0
    Not Hispanic or Latino | 6
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Per local law, ethnicity data not collected for participants located in France.
  Participants
    number analyzed (Participants) | 6
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 6
    More than one race | 0
    Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Effective Hemostasis
Description: Effective hemostasis is defined as excellent or good as assessed by the Investigator; Ineffective hemostasis is defined as moderate or poor as assessed by the Investigator. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Time Frame: Hemostasis will be assessed from the start of surgery to the end of the procedure
Population: Efficacy Set: Participants who underwent surgery and had a baseline anti-fXa activity of at least 75 nanograms (ng)/milliliter (mL) for participants receiving apixaban or rivaroxaban, 40 ng/mL for participants receiving edoxaban, and 0.25 international units (IU)/mL for participants on enoxaparin. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Measure: Count of Participants; unit: Participants
Arm/Group | Andexanet Alfa
Number analyzed (Participants) | 6
Participants | 6

2. Secondary Outcome: Percent Change From Baseline In Anti-fXa Activity To Treatment Nadir
Description: Baseline is defined as the last non-missing value on or before first study drug administration. On treatment nadir is the minimum value of anti-fXa activity during the period of time from the end of the andexanet bolus to the end of the andexanet infusion. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Time Frame: Baseline, Treatment nadir (not to exceed a total of 6.5 hours of andexanet dosing)
Population: Efficacy Set: Participants who underwent surgery and had a baseline anti-fXa activity of at least 75 ng/mL for participants receiving apixaban or rivaroxaban, 40 ng/mL for participants receiving edoxaban, and 0.25 IU/mL for participants on enoxaparin. All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Measure: Median (Full Range); unit: Percent Change
Arm/Group | Andexanet Alfa
Number analyzed (Participants) | 6
Percent Change | -96.13 [-97.4 to -89.2]

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 37
Description: All data were prespecified to be collected as a single Arm/Group for any participant who received at least 1 dose of the study drug, regardless of their dose level.
Arm/Group | Andexanet Alfa
All-Cause Mortality (participants affected / at risk) | 5/10
Serious Adverse Events (participants affected / at risk) | 7/10
Other Adverse Events (participants affected / at risk) | 2/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Andexanet Alfa (N=10)
Stress cardiomyopathy (Cardiac disorders) | 1 (1)
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 (1)
Postprocedural hematoma (Injury, poisoning and procedural complications) | 1 (1)
Ischaemic stroke (Nervous system disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Andexanet Alfa (N=10)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The study was terminated early due to the limited value as a single-arm study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-08-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT04233073/Prot_004.pdf
  • Statistical Analysis Plan (2022-04-08): https://cdn.clinicaltrials.gov/large-docs/73/NCT04233073/SAP_005.pdf